CLINICAL TRIAL: NCT06661772
Title: Influencing Factors of Vancomycin Trough Level in Critically Ill Children With Sepsis: A Single-Center Experience
Brief Title: Influencing Factors of Vancomycin Trough Level in Critically Ill Children With Sepsis
Status: Completed | Type: Observational
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Amany Mohammed El-Rebigi, MD, Lecturer of pediatric, Benha University
Other Study IDs: Rc 19-5-2024
Record Dates: First submitted 2024-10-25; First posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Critically Ill Children; Sepsis
Keywords: Vancomycin Trough Level; Sepsis; Critically ill children
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Biospecimen Retention: Samples Without DNA — Vancomycin trough levels (Human Vancomycin ELISA Kit) during treatment with at least 48 hours of PICU stay
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All pediatric Patients less than 16 years old who were diagnosed with sepsis & admitted to PICU: All consecutively hospitalized children (less than 16 years old) admitted to 30 beds in PICU who were treated with the first course of vancomycin as empirical therapy for suspected sepsis without AKI by the time of the start of treatment were enrolled in the study.
  Interventions: Diagnostic Test: Vancomycin trough concentration method

INTERVENTIONS:
Diagnostic Test: Vancomycin trough concentration method — A blood sample for VTL was drawn 30 minutes before administration, prior to the fourth dose of vancomycin, under a complete aseptic technique, unless otherwise ordered by the medical team. Vancomycin serum concentrations were measured using a Human vancomycin ELISA Kit.

SUMMARY:
The aim of the work will be to measure the vancomycin trough concentration in critically ill children with sepsis in pediatric intensive care unit and its influencing factors.

DETAILED DESCRIPTION:
Timely antibiotic administration and optimal drug dosing are crucial to achieving therapeutic antibiotic levels in critically-ill pediatric patients with suspected bacterial infection. However, drug elimination through renal excretion is often enhanced in critically ill patients . This phenomenon, referred to as augmented renal clearance (ARC), may cause sub-therapeutic serum concentrations of antibiotics through enhanced glomerular filtration, resulting in treatment failure and the generation of antibiotic-resistant strains.

Vancomycin is a tricyclic glycopeptide antibiotic with broad spectrum activity against gram-positive bacteria. It is effective for the treatment of gram positive infections and is the drug of choice for methicillin-resistant Staphylococcus aureus (MRSA). Vancomycin is poorly absorbed following oral administration. Therefore, it is commonly administered as an intravenous infusion. Approximately 50% of vancomycin is protein bound in plasma with a variable volume of distribution. An initial distribution half-life ranging from 30 min to 1 h followed by a mean terminal elimination half-life ranging from 6 h to 12 h was determined following intravenous dosing in patients with normal renal function. Metabolism is negligible and elimination occurs primarily through glomerular filtration, such that advanced renal disease substantially reduces the clearance of vancomycin resulting in an elimination half-life of about 7.5 days compared to 4-6 h in normal patients. This means that in patients with kidney failure, the dosing of vancomycin must be adjusted.

Standard treatment guidelines recommend maintaining trough levels of vancomycin between 10 and 20 mg/L. The recommended trough levels are likely to ensure optimum bactericidal activity of vancomycin, based on the minimum inhibitory concentrations (MICs) for MRSA (the lowest concentration of the drug that can prevent growth of visible bacteria).

Studies have reported a threefold increase in the risk of worsening of infections if the MICs for MRSA exceed 1.5 mg/L. However, guidelines suggest maintaining a minimum trough level of 10 mg/L for vancomycin. On the other hand, higher trough levels of vancomycin increase the risk of nephrotoxicity by two times.

Investigators have reported a correlation between serum antibiotic concentration and glomerular filtration rate (GFR). The measured GFR (mGFR), based on urine creatinine clearance over a 24-hour period, is widely used to identify patients with ARC. However, prompt administration of the proper antibiotic dose enables the serum concentration to reach therapeutic levels quickly, and the 24-hour delay when using the mGFR to identify ARC may have an adverse effect on treatment outcome in critically-ill children.

Measured glomerular filtration rate (mGFR) is often used to identify augmented renal clearance (ARC). However, in the clinical setting, estimated GFR (eGFR) is obtained more quickly and inexpensively. Therefore, eGFR can be used to identify ARC by evaluating the correlation between the eGFR and vancomycin trough level (VTL).

At our institution, empirical vancomycin therapy is commonly used due to the elevated incidence of community-acquired methicillin-resistant Staphylococcus aureus infections in the PICU. Dose adjustments based on renal function are needed, necessitating vancomycin therapeutic drug monitoring. Comparing critically ill children with sepsis to patients with normal or decreased eGFR, we hypothesize that subtherapeutic VTL has been associated with ARC.

ELIGIBILITY:
Inclusion Criteria:

* All consecutively hospitalized children (less than 16 years old), who admitted to 30 beds in PICU who were treated with the first course of vancomycin as empirical therapy for suspected sepsis without AKI by the time of the start of treatment were enrolled in the study.

Exclusion Criteria:

* children who commenced vancomycin for preventive measures, those with a history of multiple vancomycin treatment cycles, individuals showing signs of renal impairment upon initial admission to the PICU based on the pediatric risk, injury, failure, loss, end-stage renal disease (pRIFLE) criterion, and those diagnosed with congenital muscle disorders due to the potential influence of their underlying condition on serum creatinine levels.

Ages: 1 Month to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: We evaluated the influencing factors that could affect VTL in critically ill children by analyzing VTL in relation to clinical data, other laboratory investigations, dosage and frequency of vancomycin, serum creatinine concentration, CrCL, and e-GFR.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-20 (Actual)

PRIMARY OUTCOMES:
Factors affecting vancomycin trough level | 1 week
  Influencing factors that can affect Vancomycin therapeutic level

SECONDARY OUTCOMES:
Treatment failure | 1 month
  Subtherapeutic vancomycin level may lead to treatment failure

CONTACTS AND LOCATIONS:
Locations (1):
- Benha University, Cairo, Al-Qalyubia, Egypt

IPD SHARING:
Plan to Share IPD: No